CLINICAL TRIAL: NCT07018167
Title: Impact of Door-to-Needle Time on Stroke Outcomes at Gonesse Hospital
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier de Gonesse (Other)
Responsible Party: Sponsor
Other Study IDs: 0107_NEUROLOGIE
Record Dates: First submitted 2025-05-21; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Stroke; Ischemic Attack, Transient; Cerebral Infarction; Thrombolytic Therapy; Treatment Outcome
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient; Cerebral Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study looks at how quickly stroke patients receive treatment after arriving at Gonesse Hospital and whether this affects their recovery. Researchers will measure the time between a patient's arrival and the start of clot-busting treatment (called Door-to-Needle Time), as well as the time from symptom onset to hospital arrival (Home-Time). The goal is to see if treatment delays impact recovery, and to find ways to improve stroke care in the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Confirmed diagnosis of acute ischemic stroke on imaging
* Initial acute stroke care provided at Gonesse Hospital during the study period (3 months)
* Intravenous thrombolysis (r-tPA) initiated at the hospital
* Availability of clinical and timing data to calculate Door-to-Needle Time (DNT)

Exclusion Criteria:

* Patients with hemorrhagic stroke or subarachnoid hemorrhage (SAH)
* Thrombolysis initiated before hospital arrival
* Missing, incomplete, or unusable timing data for DNT calculation

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of adult patients (aged 18 and over) admitted to the Gonesse Hospital for acute ischemic stroke. All participants must have received intravenous thrombolysis (r-tPA) initiated at the hospital during the 3-month study period. Only patients with complete clinical and time-tracking data enabling the calculation of Door-to-Needle Time will be included.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Time (in minutes) from hospital arrival to thrombolysis (Door-to-Needle Time). | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- France, Gonesse, France, France